CLINICAL TRIAL: NCT05676281
Title: Healing Experiences of Adversity Among Latinos (HEALthy4You)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Family Health Centers of San Diego (Other); UCSD Center for Community Health (Unknown)
Responsible Party: Principal Investigator, Eric Hekler, Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 802492
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Stress; Childhood Obesity
Keywords: ACEs; Obesity; Adverse Childhood Experiences; 2x2 Factorial Study; Behavioral Intervention; Health Education; Healthy Together; Parenting; Protective Factors; Precision Medicine; Federally Qualified Health Centers; Latino; Hispanic; Pediatric; Whole Child Wellness
MeSH Terms: conditions — Pediatric Obesity; Obesity; Health Education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Together (includes Streetwyze) (Control/Standardized Care) (Other): Control - standardized Healthy Together program: The Healthy Together Program is not standard of care at Family Health Centers (FHC). Instead, it was originally developed by FHC clinicians interested in addressing childhood obesity and has been implemented by a limited number of clinicians at FHC. UCSD has been working in partnership with FHC to create standardized protocols and to incorporate additional research-oriented tools into this standardized protocol, which will be used as our experimental control.
  Interventions: Behavioral: Healthy Together (Control)
- Healthy Together + Promotora support (Active Comparator): In addition to the basic program described above, those randomized to this intervention will receive Promotora support. Families assigned to a promotora will receive 30-60 minutes of phone-based support weekly, with more frequent interactions that will taper starting at month 3 of the intervention. Promotoras may also provide home-visit support up to 4 times during the 6 months, based on family interest and needs. The wellness coach will try to minimize in-person meetings with FHC professionals each week and space out visits to reduce burden on families. For families in this condition, they will be asked to engage in at least 30 minutes of additional sessions per week with the promotora beyond the 1- hour allotted time working with FHC professionals.
  Interventions: Behavioral: Healthy Together + Promotora Support
- Healthy Together + Parenting training (Active Comparator): In addition to the basic program described above, those randomized to this intervention will attend Parenting Training sessions with the mental health provider at FHC. Families assigned to parenting training will receive 10-12 sessions. Sessions will focus on topics like strategies to support the child's physical, social, and emotional growth. The wellness coach will try to minimize in-person meetings with FHC professionals each week and space out visits to reduce burden on families.
  Interventions: Behavioral: Healthy Together + Parenting Training
- Healthy Togethers + Parenting Training + Promotora support (Active Comparator): Those randomized to this intervention will receive all components described above including the Healthy Together Program, Parenting Training and Promotora support. The wellness coach will try to minimize in-person meetings with FHC professionals each week and space out visits to reduce burden on families.. Families in this group will also be asked to engage in at least 30-60 minutes of additional sessions per week including up to 4 home visits.
  Interventions: Behavioral: Healthy Togethers + Parenting Training + Promotora support

INTERVENTIONS:
Behavioral: Healthy Together (Control) — The total number of sessions families will engage with will be negotiated between the Families and their Care providers. This allows for families to receive care while still honoring their constraints, such as the amount of time they can dedicate per week and over the course of the study, to the intervention. The maximum number of possible sessions include:
  * 6 Sessions with a Wellness Coach
  * 4-8 sessions with a Dietician
  * 4-8 sessions of Physical Theraphy
  * 1 session during month 1 or 2 Streetwyze Training
  * Safety Net Referrals
  Arms: Healthy Together (includes Streetwyze) (Control/Standardized Care)
Behavioral: Healthy Together + Promotora Support — The total number of sessions families will engage with will be negotiated between the Families and their Care providers. This allows for families to receive care while still honoring their constraints, such as the amount of time they can dedicate per week and over the course of the study, to the intervention. The maximum number of possible sessions include:
  * 6 Sessions with a Wellness Coach
  * 4-8 sessions with a Dietician
  * 4-8 sessions of Physical Theraphy
  * 1 session during month 1 or 2 Streetwyze Training
  * Safety Net Referrals
  * 16-20 Promotora (in home case management) Sessions (weekly first 2 months, afterwards at least bi-weekly)
  Arms: Healthy Together + Promotora support
Behavioral: Healthy Together + Parenting Training — The total number of sessions families will engage with will be negotiated between the Families and their Care providers. This allows for families to receive care while still honoring their constraints, such as the amount of time they can dedicate per week and over the course of the study, to the intervention. The maximum number of possible sessions include:
  * 6 Sessions with a Wellness Coach
  * 4-8 sessions with a Dietician
  * 4-8 sessions of Physical Theraphy
  * 1 session during month 1 or 2 Streetwyze Training
  * Safety Net Referrals
  * 6-10 Parenting Sessions with a Family Health Centers Mental Health Provider using the Incredible Years Curriculum
  Arms: Healthy Together + Parenting training
Behavioral: Healthy Togethers + Parenting Training + Promotora support — The total number of sessions families will engage with will be negotiated between the Families and their Care providers. This allows for families to receive care while still honoring their constraints, such as the amount of time they can dedicate per week and over the course of the study, to the intervention. The maximum number of possible sessions include:
  * 6 Sessions with a Wellness Coach
  * 4-8 sessions with a Dietician
  * 4-8 sessions of Physical Theraphy
  * 1 session during month 1 or 2 Streetwyze Training
  * Safety Net Referrals
  * 16-20 Promotora (in home case management) Sessions (weekly first 2 months, afterwards at least bi-weekly)
  * 8-10 Parenting Sessions with a Family Health Centers Mental Health Provider using the Incredible Years Curriculum
  Arms: Healthy Togethers + Parenting Training + Promotora support

SUMMARY:
Healing Experiences of Adversity Among Latinos (HEALthy4You) is a project funded by the California Initiative for the Advancement of Precision Medicine ("Advancing a Precision Population Health Approach to ACEs to Reduce Health Disparities"). The long-term goal of this project is to develop community-centered, culturally Appropriate, precision Interventions that can be delivered within Federally Qualified Healthcare Centers (FQHCs) for Latino Families, to reduce Adverse Child Events (ACES) risks and treat childhood obesity. UCSD in conjunction with Family Health Centers of San Diego (FHCSD) will conduct a 2x2 factorial trial with four groups meant to determine what combination of intervention components influence family protective factors (a key marker for reduced risk of the deleterious effects of systemic and family/individual stressors that are a critical part of ACEs) and childhood obesity.

ELIGIBILITY:
Inclusion Criteria:

* Child
* Currently a patient at Family Health Centers of San Diego
* Age 5-11 years old
* BMI ≥ 85th percentile to 99.9th percentile
* Social determination or risk for ACE determined as being a patient receiving care at an FQHC (confirmed via provider)
* Parent
* Parent or guardian (including non-biological parent or relative) willing to participate
* Self-identification as Hispanic or Latino
* 18 years or older
* English or Spanish speaking
* Willingness to commit to 6 months of the program

Exclusion Criteria:

* Serious Developmental Disability (parent or child)
* Serious Mental Health Illness (parent or child)

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Parents' Assessment of Protective Factors Self-Report Scale (comparison baseline to 6-months) | 6 months
  Parents' Assessment of Protective Factors (PAPF) Instrument consists of 36 items to measure the presence, strength, and growth of parents' self-reported beliefs, feelings, and behaviors that are regarded as indicators of the Strengthening Families protective factors using a 5-point response system from "Not at all like me" to "Very much like me" (Score scale: 0 Low - 3.99 High)

SECONDARY OUTCOMES:
Changes to Child Body Mass Index (BMI) from baseline to 6 months | 6 months
  Weight and height will be combined to report BMI in kg/m^2.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Family Health Centers of San Diego, San Diego, California
  - Jessica Chapman, San Diego, California